CLINICAL TRIAL: NCT01380132
Title: Safety and Efficacy of Anorectal Application of Dx-gel for Treatment of Anal Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Olof Nilsson, Uppsala university
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nasha Dx Pilot study; 03 464 (Other: EPN Uppsala)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-02

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Treatment; Surgery
MeSH Terms: conditions — Fecal Incontinence | interventions — dextranomer-hyaluronic acid copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anal injection of Nasha Dx (Experimental)
  Interventions: Procedure: Anal injection of Nasha Dx

INTERVENTIONS:
Procedure: Anal injection of Nasha Dx — Submucous injection of Nasha Dx 5-10 mm above dentate line
  Other Names: Solesta

SUMMARY:
The purpose of this study is to determine whether anorectal application of Nasha Dx is safe and effective for treatment of anal incontinence.

DETAILED DESCRIPTION:
Patients not fully improved after 1:st injection were offered reinjection after 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Incontinence to loose or solid stool at least once weekly (Millers incontinence score 6-12).
* Age 18-80
* Available for follow-up for the duration of the study
* Written informed consent.

Exclusion Criteria:

* Sphincter defect visible on anal ultrasound.
* Pregnancy.
* Rectal prolapse or inflammatory bowel disease.
* Recent (within 6 months) anal surgery except for haemorrhoids.
* Anorectal sepsis.
* Anticoagulant medication or bleeding diathesis.

Ages: 18 Years to 80 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-02; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Treatment response as measured by a 50% reduction in no of incontinence episodes. | One year posttreatment

SECONDARY OUTCOMES:
Adverse events | One year posttreatment
Global assessment | One year posttreatment
  Graded by the patient as excellent, good, fair or poor
Change in incontinence episodes | One year posttreatment
  Measured relative baseline based on a 4-week diary
Quality of life | One year posttreatment
  Measured with a validated bowel function questionnaire
Adverse events | Two years posttreatment
Global assessment | Two years posttreatment
  Graded by the patient as excellent, good, fair or poor
Change in incontinence episodes | Two years posttreatment
  Measured relative baseline based on a 4-week diary
Quality of life | Two years posttreatment
  Measured with a validated bowel function questionnaire
Treatment response as measured by a 50% reduction in no of incontinence episodes. | Two years posttreatment

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm JR Graf, Prof., Principal Investigator — Inst of Surgical Sciences, Uppsala university
Locations (1):
- Department of Surgery, University Hospital, 751 82 Uppsala, Sweden

REFERENCES:
- [Result] Danielson J, Karlbom U, Sonesson AC, Wester T, Graf W. Submucosal injection of stabilized nonanimal hyaluronic acid with dextranomer: a new treatment option for fecal incontinence. Dis Colon Rectum. 2009 Jun;52(6):1101-6. doi: 10.1007/DCR.0b013e31819f5cbf. PMID 19581853